CLINICAL TRIAL: NCT06497517
Title: A Phase 1, Single Center, Single Dose, Open-Label, Randomized, 2-Way Crossover Study to Investigate the Food Effect on the Pharmacokinetics of Camlipixant in Healthy Male and Female Participants
Brief Title: A Study to Investigate the Effect of Food on Camlipixant Concentrations in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bellus Health Inc. - a GSK company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 222708
Record Dates: First submitted 2024-07-05; First posted 2024-07-11 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Cough
Keywords: Camlipixant; GSK5464714-camlipixant; Healthy Participants; Pharmacokinetics; Cross-over Study
MeSH Terms: conditions — Cough

STUDY DESIGN:
Masking Description: This is an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequence 1 (Experimental): In sequence 1, eligible participants will be randomly assigned to 1 of 2 sequences to receive single dose of GSK5464714- Camlipixant on Day 1 under fasting condition (Treatment A), followed by single dose of GSK5464714 in fed condition (Treatment B). There will be a washout period of minimum 7 days between each period.
  Interventions: Drug: GSK5464714- Camlipixant
- Sequence 2 (Experimental): In sequence 2, eligible participants will be randomly assigned to 1 of 2 sequences to receive single dose of GSK5464714- Camlipixant on Day 1 in fed condition (Treatment B), followed by single dose of GSK5464714 under fasting condition (Treatment A). There will be a washout period of minimum 7 days between each period.
  Interventions: Drug: GSK5464714- Camlipixant

INTERVENTIONS:
Drug: GSK5464714- Camlipixant — GSK5464714- Camlipixant will be administered
  Other Names: Camlipixant

SUMMARY:
This study is a single center, single dose, open-label, randomly assigned 2-way crossover study. The study will investigate the food effect on the pharmacokinetics of Camlipixant (GSK5464714) in healthy male and female participants. Eligible participants will be randomized to pre-defined sequences. There will be a washout of minimum 7 days between each dose of treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, clinical laboratory tests, vital sign measurements, and 12-lead ECGs including the following:

  * Seated blood pressure (after 5 mins), average of 3 readings, is greater than or equal to (>=) 90/55 millimetre of mercury (mmHg) and less than or equal (<=)140/90 mmHg at the screening visit.
  * Seated heart rate, average of 3 readings, is >= 40 beats per minutes (bpm) and <= 99 bpm at the screening visit.
  * Corrected QT interval using the Fridericia formula (QTcF) on ECG, average of 3 readings, is <= 450 millisecond (msec) and 12-lead ECG findings considered normal or not clinically significant by the investigator or designee at the screening visit.
* Aspartate transferase (AST), Alanine transaminase (ALT), direct bilirubin, indirect bilirubin, and total bilirubin within normal ranges at the screening visit and check-in. Only abnormal values up to 1.5 x upper limit of normal may be repeated once
* Continuous non-smoker who has never used nicotine- or tobacco-containing products or light smoker for the last 6 months prior to study screening
* Body weight ≥ 50.0 kilogram (kg) and Body mass index (BMI) within the range 18.5 to 32.0 kilogram per meter square (kg/m2) (inclusive) at Screening.
* Male and female participants must follow protocol-specified contraception guidance.
* Female participants: A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies

  * Is a woman of nonchildbearing potential (WONCBP)
  * Is a Woman of childbearing potential (WOCBP) and using a contraceptive method that is highly effective
  * A WOCBP must have a negative highly sensitive serum pregnancy test within 24 hours before the first dose of study intervention (i.e., Day -1 of each treatment period)
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.
* Must be willing and able to comply with the protocol.

Exclusion Criteria:

* History or presence of clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, biliary (including gallstones or previous cholecystectomy), endocrine, hematologic, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention or interfering with the interpretation of data.
* Have a history of malignant neoplasm (excepting definitively treated non melanoma skin cancer or carcinoma in situ of the uterine cervix, which may be enrolled at any time) within the last 5 years.
* Past or intended use of over-the-counter or prescription medication including herbal medications within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to dosing.
* Participation in the clinical study would result in loss of blood or blood products in excess of 500 milliliter (mL) within 3 months.
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
* Current enrolment or past participation in another investigational clinical study in which an investigational intervention (e.g., drug, vaccine, invasive device) was administered within the last 30 days or 5.5 half-lives before signing of consent in any other clinical study involving an investigational study intervention or any other type of medical research.
* Current enrolment or past participation in this clinical study.
* Positive pre-study drug/alcohol screen, including tetrahydrocannabinol.
* Positive Human immunodeficiency virus (HIV) antibody test.
* Positive coronavirus (severe acute respiratory syndrome coronavirus 2 [SARS-CoV-2]) polymerase chain reaction test at check-in.
* Presence of Hepatitis B surface antigen (HBsAg) or Hepatitis B core antibody (HBcAb) at screening or within 3 months prior to first dose of study intervention.
* Positive Hepatitis C virus (HCV) antibody test result at screening or within 3 months prior to starting study intervention.
* Total bilirubin >1.5x upper limit of normal (ULN), including participants with Gilbert's syndrome.
* Regular alcohol consumption within 6 months prior to the clinical study defined as: For sites in United States of America (USA), an average weekly intake of 3 units for males or 1.5 units for females.
* History of known drugs of abuse, including tetrahydrocannabinol, in last 5 years.
* Sensitivity to heparin or heparin-induced thrombocytopenia.
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the clinical study.
* Use of any products intended to treat medical conditions that are not approved by the governing health authority in a given country or region (for example, herbal medicine, health supplements, traditional medicine, homeopathic remedies, etc.), within past 30 days prior to signing the consent and during the study.
* Any dietary restrictions that would prevent the participant from consuming the site menu/meals.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2024-07-09 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2024-08-26 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve (AUC) from Time Zero to Infinity Post-Dose [AUC(0-inf) | Up to Day 3 for each period
Maximum Observed Plasma Drug Concentration (Cmax) | Up to Day 3 for each period

SECONDARY OUTCOMES:
Time to Maximum Observed Plasma Drug Concentration (Tmax) | Up to Day 3 for each period
Apparent Terminal Phase Half-Life (t½) | Up to Day 3 for each period
Apparent Oral Clearance (CL/F) | Up to Day 3 for each period
AUC from Time Zero to Last Quantifiable Concentration [AUC(0-t) | Up to Day 3 for each period
Apparent Volume of Distribution (Vz/F) | Up to Day 3 for each period
Number of Participants Reported for Adverse events, Serious Adverse Events and Adverse Events of Special Interest | Up to 3 weeks
Absolute Values for Clinical Laboratory Parameters Over Time | Up to 3 weeks
Absolute Values for 12- Lead Electrocardiogram (ECG) Over Time | Up to 3 weeks
Absolute Values for Vital Sign Measurements Over Time | Up to 3 weeks
Changes from Baseline for Clinical Laboratory Parameters Over Time | Up to 3 weeks
Changes from Baseline for 12- Lead ECG Over Time | Up to 3 weeks
Changes from Baseline for Vital Sign Measurements Over Time | Up to 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/